CLINICAL TRIAL: NCT04549636
Title: Prospective Longitudinal Study to Characterize and Understand the Clinical Relevance of SARS-CoV2 Related Ventilation and Perfusion Injury Evaluated by V/Q SPECT-CT in an Asthmatic and Healthy Population
Brief Title: COVID-19 Related Lung Ventilation and Perfusion Injury
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: FIRH002
Record Dates: First submitted 2020-08-28; First posted 2020-09-16 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Covid-19; Asthma; Healthy
Keywords: covid-19; lung ventilation; lung perfusion; V/Q SPECT; lung health; Technegas
MeSH Terms: conditions — COVID-19; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- healthy COVID-19+: Individuals who recently recovered from COVID-19 and who have no history of lung disease
  Interventions: Other: V/Q SPECT-CT; Other: St. George's Respiratory Questionnaire (SGRQ); Other: mMRC (Modified Medical Research Council) Dyspnea Scale; Other: Six-minute walk test (6MWT); Other: Spirometry; Other: Plethysmography & DLCO; Other: Airwave Oscillometry
- asthmatic COVID-19+: Individuals who recently recovered from COVID-19 and who have asthma
  Interventions: Other: V/Q SPECT-CT; Other: St. George's Respiratory Questionnaire (SGRQ); Other: mMRC (Modified Medical Research Council) Dyspnea Scale; Other: Six-minute walk test (6MWT); Other: Spirometry; Other: Plethysmography & DLCO; Other: Airwave Oscillometry
- healthy COVID-19-: Individuals who have not been diagnosed with COVID-19 and who have no history of lung disease
  Interventions: Other: V/Q SPECT-CT; Other: St. George's Respiratory Questionnaire (SGRQ); Other: mMRC (Modified Medical Research Council) Dyspnea Scale; Other: Six-minute walk test (6MWT); Other: Spirometry; Other: Plethysmography & DLCO; Other: Airwave Oscillometry
- asthmatic COVID-19-: Individuals who have not been diagnosed with COVID-19 and who have asthma
  Interventions: Other: V/Q SPECT-CT; Other: St. George's Respiratory Questionnaire (SGRQ); Other: mMRC (Modified Medical Research Council) Dyspnea Scale; Other: Six-minute walk test (6MWT); Other: Spirometry; Other: Plethysmography & DLCO; Other: Airwave Oscillometry

INTERVENTIONS:
Other: V/Q SPECT-CT — At visits 1 and 2, ventilation will be assessed by 99mTc Technegas SPECT ventilation scan and perfusion will be assessed by 99mTc Macroaggregated Albumin SPECT perfusion scan.
Other: St. George's Respiratory Questionnaire (SGRQ) — At visits 1 and 2, quality of life will be evaluated using the St. George's Respiratory Questionnaire (SGRQ).
Other: mMRC (Modified Medical Research Council) Dyspnea Scale — At visits 1 and 2, dyspnea will be evaluated using the mMRC (Modified Medical Research Council) Dyspnea Scale.
Other: Six-minute walk test (6MWT) — At visits 1 and 2, exercise capacity will be evaluated using the six-minute walk test (6MWT).
Other: Spirometry — At visits 1 and 2, spirometry will be performed to quantify the forced expiratory volume in one second (FEV1), the forced vital capacity (FVC) and FEV1/FVC.
Other: Plethysmography & DLCO — At visits 1 and 2, plethysmography and the diffusing capacity of the lung for carbon monoxide (DLCO) will be performed.
Other: Airwave Oscillometry — At visits 1 and 2, airwave oscillometry will be performed to obtain resistance (R) and reactance (X) at 5 Hz (R5) and 19 Hz (R19). The resonance frequency (fres), area above the reactance curve (AX) and the heterogeneity of obstruction (R5-19) will be derived from R and X.

SUMMARY:
Little is currently known about the immediate and long-term effect of COVID-19 on lung ventilation (delivery of air to the lungs) and lung perfusion (delivery of blood to the lungs). Some people who survive COVID-19 may have lung ventilation and/or perfusion injury that persists following COVID-19 recovery. This lung injury may be related to inflammation in the lung, breathlessness, exercise limitation and reduced quality of life. Therefore, towards the goal of understanding the effects of COVID-19 on lung health, the purpose of this study is to characterize and understand the clinical relevance of COVID-19 related lung ventilation and perfusion injury and associated inflammatory status, ≤4 weeks and 6-months following COVID-19 recovery in an asthmatic and healthy population. To do this, an asthmatic and healthy population who have, and have not, been previously diagnosed with COVID-19 will be studied.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Males and females ≥ 18 years of age
* Individuals able and willing to provide written informed consent
* Individuals able and willing to comply with the study protocol

For participants with asthma:

* Individuals with physician confirmed asthma (12% bronchodilator reversibility or PC20 methacholine less than 8mg/ml)
* Individuals treated with inhaled corticosteroids, oral corticosteroids and/or anti-T2 biologics

For participants who recently recovered from covid-19:

* Individuals previously diagnosed with covid-19 confirmed by FLOQswab test
* Individuals who recently (≤4-weeks) recovered from covid-19

Exclusion Criteria:

For all participants:

* Males and females < 18 years of age
* Individuals who are unable to read and/or understand English
* Individuals who are pregnant or breastfeeding
* Individuals who currently smoke or are an ex-smoker with ≥10 pack-year smoking history
* Individuals who in the opinion of the investigator, are mentally or legally incapacitated, preventing informed consent from being obtained
* Individuals who are unable to complete one or more study manoeuvres

For participants with no history of lung disease:

* Individuals with a history of respiratory infection or disease

For participants who have not been diagnosed with covid-19:

* Individuals who have previously had covid-19 confirmed by FLOQswab test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Short-term difference in ventilation defect percent assessed by ventilation SPECT-CT - healthy | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung ventilation between healthyCOVID-19+ and healthyCOVID-19- participants
Short-term difference in perfusion defect percent assessed by perfusion SPECT-CT - healthy | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung perfusion between healthyCOVID-19+ and healthyCOVID-19- participants
Short-term difference in lung ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - healthy | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung ventilation/perfusion mismatch between healthyCOVID-19+ and healthyCOVID-19- participants
Long-term difference in ventilation defect percent assessed by ventilation SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung ventilation between healthyCOVID-19+ and healthyCOVID-19- participants
Long-term difference in perfusion defect percent assessed by perfusion SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung perfusion between healthyCOVID-19+ and healthyCOVID-19- participants
Long-term difference in ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung ventilation/perfusion mismatch between healthyCOVID-19+ and healthyCOVID-19- participants
Short-term difference in ventilation defect percent assessed by ventilation SPECT-CT - asthmatic | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung ventilation between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Short-term difference in perfusion defect percent assessed by perfusion SPECT-CT - asthmatic | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung perfusion between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Short-term difference in ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - asthmatic | ≤4-weeks post COVID-19 recovery (Visit 1)
  The short-term difference in lung ventilation/perfusion mismatch between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Long-term difference in ventilation defect percent assessed by ventilation SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung ventilation between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Long-term difference in perfusion defect percent assessed by perfusion SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung perfusion between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Long-term difference in ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  The long-term difference in lung ventilation/perfusion mismatch between asthmaticCOVID-19+ and asthmaticCOVID-19- participants
Longitudinal change in ventilation defect percent assessed by ventilation SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung ventilation between healthyCOVID-19+ and healthyCOVID-19- participants
Longitudinal change in perfusion defect percent assessed by perfusion SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung perfusion between healthyCOVID-19+ and healthyCOVID-19- participants
Longitudinal change in ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - healthy | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung ventilation/perfusion mismatch between healthyCOVID-19+ and healthyCOVID-19- participants
Longitudinal change in ventilation defect percent assessed by ventilation SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung ventilation between asthmaticCOVID-19+ and asthmaticCOVID-19- participants.
Longitudinal change in perfusion defect percent assessed by perfusion SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung perfusion between asthmaticCOVID-19+ and asthmaticCOVID-19- participants.
Longitudinal change in ventilation/perfusion mismatch assessed by ventilation/perfusion SPECT-CT - asthmatic | 6-months post COVID-19 recovery (Visit 2)
  Difference in the 6-month change in lung ventilation/perfusion mismatch between asthmaticCOVID-19+ and asthmaticCOVID-19- participants.

SECONDARY OUTCOMES:
Correlation of lung ventilation with the St. George's Respiratory Questionnaire (SGRQ) score ≤4-weeks post COVID-19 recovery | ≤4-weeks post COVID-19 recovery (Visit 1)
  In COVID-19+ participants, the correlation of lung ventilation with the St. George's Respiratory Questionnaire (SGRQ) score ≤4-weeks post COVID-19 recovery (Visit 1).
Correlation of lung ventilation with six-minute walk distance (6MWD) ≤4-weeks post COVID-19 recovery | ≤4-weeks post COVID-19 recovery (Visit 1)
  In COVID-19+ participants, the correlation of lung ventilation with six-minute walk distance (6MWD) ≤4-weeks post COVID-19 recovery (Visit 1).
Correlation of lung ventilation with the forced expiratory volume in one second (FEV1) ≤4-weeks post COVID-19 recovery | ≤4-weeks post COVID-19 recovery (Visit 1)
  In COVID-19+ participants, the correlation of lung ventilation with the forced expiratory volume in one second (FEV1) ≤4-weeks post COVID-19 recovery (Visit 1).
Correlation of lung ventilation with the diffusing capacity of the lung for carbon monoxide (DLCO) ≤4-weeks post COVID-19 recovery | ≤4-weeks post COVID-19 recovery (Visit 1)
  In COVID-19+ participants, the correlation of lung ventilation with the diffusing capacity of the lung for carbon monoxide (DLCO) ≤4-weeks post COVID-19 recovery (Visit 1).
Correlation of lung ventilation with the St. George's Respiratory Questionnaire (SGRQ) score 6-months post COVID-19 recovery | 6-months post COVID-19 recovery (Visit 2)
  In COVID-19+ participants, the correlation of lung ventilation with the St. George's Respiratory Questionnaire (SGRQ) score 6-months post COVID-19 recovery (Visit 2).
Correlation of lung ventilation with six-minute walk distance (6MWD) 6-months post COVID-19 recovery | 6-months post COVID-19 recovery (Visit 2)
  In COVID-19+ participants, the correlation of lung ventilation with six-minute walk distance (6MWD) 6-months post COVID-19 recovery (Visit 2).
Correlation of lung ventilation with the forced expiratory volume in one second (FEV1) 6-months post COVID-19 recovery | 6-months post COVID-19 recovery (Visit 2)
  In COVID-19+ participants, the correlation of lung ventilation with the forced expiratory volume in one second (FEV1) 6-months post COVID-19 recovery (Visit 2).
Correlation of lung ventilation with the diffusing capacity of the lung for carbon monoxide (DLCO) 6-months post COVID-19 recovery | 6-months post COVID-19 recovery (Visit 2)
  In COVID-19+ participants, the correlation of lung ventilation with the diffusing capacity of the lung for carbon monoxide (DLCO) 6-months post COVID-19 recovery (Visit 2).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Svenningsen, PhD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.